CLINICAL TRIAL: NCT01206127
Title: DSAEK- Postoperative Positioning and Transplant Dislocation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Prof. Liv Drolsum, MD, PhD, Department of Ophthalmology, Oslo University Hospital Ullevål, Norway
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 239-08/344c(REK)-1
Record Dates: First submitted 2010-09-20; First posted 2010-09-21 (Estimated); Last update posted 2010-09-21 (Estimated); Status verified 2010-09

CONDITIONS: Corneal Transplantation; Descemet Stripping Automated Endothelial Keratoplasty; Fuchs' Endothelial Dystrophy; Corneal Dystrophies, Hereditary
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy; Corneal Dystrophies, Hereditary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Postoperative positioning: Bed rest (Other): Patients in this group must be lying down facing up 2 hours postoperatively
  Interventions: Other: Postoperative positioning: Bed rest
- Postoperative positioning: Sitting up (Other): Patients in this group should be sitting up in a chair 2 hours postoperatively
  Interventions: Other: Postoperative positioning: Sitting up

INTERVENTIONS:
Other: Postoperative positioning: Bed rest — Patients in this group should be lying down facing up 2 hours postoperatively
  Arms: Postoperative positioning: Bed rest
Other: Postoperative positioning: Sitting up — Patients in this group should be sitting up in a chair 2 hours postoperative
  Arms: Postoperative positioning: Sitting up

SUMMARY:
Corneal transplant is a surgical procedure where a damaged or diseased cornea is replaced by donated corneal tissue (the graft) in its entirety (penetrating keratoplasty) or in part (lamellar keratoplasty). One type of lamellar keratoplasty is DSAEK (Descemet's Stripping Automated Endothelial Keratoplasty), where only the damaged posterior section of the cornea is replaced.

The purpose of this study is to investigate how immediate postoperative positioning of the patient affects the dislocation rate of the corneal graft. Since this is a new surgical method, little scientific documentation has been published in this area.

DETAILED DESCRIPTION:
Corneal transplant is a surgical procedure where a damaged or diseased cornea is replaced by donated corneal tissue (the graft) in its entirety (penetrating keratoplasty) or in part (lamellar keratoplasty). One type of lamellar keratoplasty is DSAEK (Descemet's Stripping Automated Endothelial Keratoplasty), where only the damaged posterior section of the cornea is replaced.

To get the graft in the right position inside the eyes anterior chamber, the anterior chamber is fully filled with air, and the patient is placed in a supine position looking facing up for different amount of time depending on the surgeon. In this way the air bubble will press the graft in the right position and prevent dislocation. Our experience is that since the anterior chamber of the eye already is fully filled with air, it does not matter how the patient is positioned postoperatively regarding graft dislocation.

Our hypothesis is that the immediate postoperative positioning is insignificant. If this can be significantly proved this may enhance the patients comfort postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Corneal dystrophy requiring corneal transplantation
* Patients written permission
* Pseudophakia

Exclusion Criteria:

* Uncontrolled glaucoma
* Phakia or aphakia
* Shallow anterior chamber
* Fibrotic cornea
* Demented patients
* Claustrophobic patients
* Patients that do not want to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-09; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Graft dislocation measured by slit lamp examination | 5 years
  Graft dislocation is checked 2 hours postoperatively, they day after the surgery, 1 week after, 1 month, and then every 3. month for 1 year, and then every 6. months for 5 years.

SECONDARY OUTCOMES:
Intraocular pressure (IOP) | 5 years
  The intraocular pressure (IOP) is measured at every postoperative control
Visual Acuity | 5 years
  Visual Acuity is measured at every postoperative control
Endothelial cell count of the graft | 5 years
  Endothelial cell count of the graft is measured at every postoperative control

CONTACTS AND LOCATIONS:
Overall Officials: Liv Drolsum, Prof.,MD,PhD, Study Director — Department of Ophthalmology, Oslo University Hospital, Norway
Locations (1):
- Departement of Ophthalmology, Oslo University Hospital, Norway, Oslo, Oslo County, Norway

REFERENCES:
- [Background] Price MO, Gorovoy M, Benetz BA, Price FW Jr, Menegay HJ, Debanne SM, Lass JH. Descemet's stripping automated endothelial keratoplasty outcomes compared with penetrating keratoplasty from the Cornea Donor Study. Ophthalmology. 2010 Mar;117(3):438-44. doi: 10.1016/j.ophtha.2009.07.036. Epub 2010 Jan 19. PMID 20031230
- [Background] Price MO, Giebel AW, Fairchild KM, Price FW Jr. Descemet's membrane endothelial keratoplasty: prospective multicenter study of visual and refractive outcomes and endothelial survival. Ophthalmology. 2009 Dec;116(12):2361-8. doi: 10.1016/j.ophtha.2009.07.010. Epub 2009 Oct 28. PMID 19875170
- [Background] Dapena I, Ham L, Melles GR. Endothelial keratoplasty: DSEK/DSAEK or DMEK--the thinner the better? Curr Opin Ophthalmol. 2009 Jul;20(4):299-307. doi: 10.1097/ICU.0b013e32832b8d18. PMID 19417653